CLINICAL TRIAL: NCT03731039
Title: Survey of Postoperative Pain Control in Adults After Different Types of Surgeries.
Brief Title: Postoperative Pain in Adult Patients.
Status: Completed | Type: Observational
Sponsor: Andrzej Frycz Modrzewski Krakow University (Other)
Responsible Party: Principal Investigator, Lucyna Tomaszek, PhD, Specialist Nurse in Anesthesia and Intensive Care, Andrzej Frycz Modrzewski Krakow University
Other Study IDs: WLNZ/DS/3/2018
Record Dates: First submitted 2018-11-02; First posted 2018-11-06 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Pain, Postoperative; Surgical Procedures, Operative
Keywords: Postoperative pain; Anxiety; Depression; Adult
MeSH Terms: conditions — Pain, Postoperative; Anxiety Disorders; Depression | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- SURGICAL PROCEDURES ASSOCIATED WITH SLIGHT TISSUE DAMAGE
  Interventions: Other: Observational study
- SURGICAL PROCEDURES ASSOCIATED WITH MODERATE TISSUE DAMAGE
  Interventions: Other: Observational study
- SURGICAL PROCEDURES ASSOCIATED WITH SUBSTANTIAL TISSUE DAMAGE
  Interventions: Other: Observational study

INTERVENTIONS:
Other: Observational study — Pain assessment, Anxiety assessment, Depression assessment

SUMMARY:
Each surgical intervention associated with even a minor tissue injury is a source of pain which needs to be effectively controlled. Although the Polish national guidelines for post-operative pain management have been published, many patients experience moderate and severe pain in the postoperative period. The aim of this study is (1) to assess pain severity among adult patients after different types of surgeries; (2) to identify demographic and clinical factors associated with postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* adult
* elective surgery
* the American Society of Anesthesiologists score 1-3

Exclusion Criteria:

* diagnosed mental illness, alcohol abuse disorders, intellectual disability
* traumatic events within the last 6 months (e.g. death, breakdown of a relationship, job loss)
* problems with verbal communication

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients underoing surgical procedures performed on general or regional anesthesia.
Sampling Method: Probability Sample
Enrollment: 620 (Actual)
Dates: Start 2017-09-21 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Pain intensity scores at rest | first 24 hours after surgery
  Pain intensity is assessed using the Numeric Rating Scale (NRS), where 0 meant no pain and 10 maximum pain. Numeric scores of 1-3, 4-6, and 7-10 corresponded to mild, moderate and severe pain.
Pain intensity scores on movement | first 24 hours after surgery
  Pain intensity is assessed using the Numeric Rating Scale (NRS), where 0 meant no pain and 10 maximum pain. Numeric scores of 1-3, 4-6, and 7-10 corresponded to mild, moderate and severe pain.

SECONDARY OUTCOMES:
Anxiety scores | day prior to surgery
  Anxiety is evaluated using the Hospital Anxiety and Depression Scale - HADS. It consists of 7 items grouped in sub-scales: anxiety (HADS-A) and depression (HADS-D). The answers describe the patient's well-being over the last week and are coded on a scale of 0-3 points.
  HADS-A: the total score amounts to 0-21 points (0-7 points = norm, 8-10 = borderline, ≥11 points = clinical levels of symptoms).
Depression scores | day prior to surgery
  Depression is evaluated using the Hospital Anxiety and Depression Scale - HADS. It consists of 7 items grouped in sub-scales: anxiety (HADS-A) and depression (HADS-D). The answers describe the patient's well-being over the last week and are coded on a scale of 0-3 points.
  HADS-D: the total score amounts to 0-21 points (0-7 points = norm, 8-10 = borderline, ≥11 points = clinical levels of symptoms).

CONTACTS AND LOCATIONS:
Overall Officials: Lucyna Tomaszek, Study Director — Andrzej Frycz Modrzewski Krakow University
Locations (1):
- Andrzej Frycz-Modrzewski Krakow University, Krakow, Lesser Poland Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Borys M, Zyzak K, Hanych A, Domagala M, Galkin P, Galaszkiewicz K, Klaput A, Wroblewski K, Miekina J, Onichimowski D, Czuczwar M. Survey of postoperative pain control in different types of hospitals: a multicenter observational study. BMC Anesthesiol. 2018 Jul 18;18(1):83. doi: 10.1186/s12871-018-0551-3. PMID 30021520
- [Background] Misiolek H, Cettler M, Woron J, Wordliczek J, Dobrogowski J, Mayzner-Zawadzka E. The 2014 guidelines for post-operative pain management. Anaesthesiol Intensive Ther. 2014 Sep-Oct;46(4):221-44. doi: 10.5603/AIT.2014.0041. No abstract available. PMID 25293474
- [Result] Tomaszek L, Debska G. Knowledge, compliance with good clinical practices and barriers to effective control of postoperative pain among nurses from hospitals with and without a "Hospital without Pain" certificate. J Clin Nurs. 2018 Apr;27(7-8):1641-1652. doi: 10.1111/jocn.14215. Epub 2018 Mar 2. PMID 29218814